CLINICAL TRIAL: NCT00000973
Title: Pyrimethamine Pharmacokinetics in HIV Positive Patients Seropositive for Toxoplasma Gondii
Brief Title: A Study of Pyrimethamine in the Treatment of Infection by a Certain Parasite in HIV-Positive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 102; 11077 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Toxoplasmosis, Cerebral; HIV Infections
Keywords: Toxoplasmosis; Toxoplasma; Pyrimethamine; Leucovorin; Drug Evaluation; Encephalitis; Zidovudine
MeSH Terms: conditions — Toxoplasmosis, Cerebral; HIV Infections; Toxoplasmosis; Encephalitis | interventions — Pyrimethamine; Leucovorin; Zidovudine

INTERVENTIONS:
Drug: Pyrimethamine
Drug: Leucovorin calcium
Drug: Zidovudine

SUMMARY:
To determine the manner in which pyrimethamine is metabolized and excreted in patients currently receiving zidovudine (AZT). An important goal of this measurement is to establish the optimal dose of pyrimethamine necessary to prevent the development of toxoplasmosis in AIDS patients or delay the subsequent return of toxoplasmic encephalitis.

Encephalitis caused by Toxoplasma gondii has emerged as the most frequent cause of focal central nervous system infection in patients with AIDS. Untreated, the encephalitis is fatal. The best treatment for this disease has not been determined. Presently it is standard practice to administer a combination of pyrimethamine and sulfadiazine. Little is known about the pharmacokinetics of pyrimethamine in patients with AIDS receiving AZT. Furthermore, there are reports that patients already exposed to toxoplasmosis may not have uniform absorption of pyrimethamine.

DETAILED DESCRIPTION:
Encephalitis caused by Toxoplasma gondii has emerged as the most frequent cause of focal central nervous system infection in patients with AIDS. Untreated, the encephalitis is fatal. The best treatment for this disease has not been determined. Presently it is standard practice to administer a combination of pyrimethamine and sulfadiazine. Little is known about the pharmacokinetics of pyrimethamine in patients with AIDS receiving AZT. Furthermore, there are reports that patients already exposed to toxoplasmosis may not have uniform absorption of pyrimethamine.

Patients receive the study treatment for a total of 22 days. Patients are given an initial dose of pyrimethamine followed by a lower dose given as a single oral daily dose for 21 days. Patients continue to receive AZT at the dose prescribed prior to enrollment in the study. Patients receive leucovorin calcium once a day. Neither the leucovorin calcium nor the AZT are provided through the study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine for Pneumocystis carinii pneumonia prophylaxis.
* Isoniazid not initiated during study period.
* Methadone maintenance.

Required:

* Stable prescribed dose of zidovudine (AZT) of at least 500 mg/day.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Prior history of toxoplasmic encephalitis.
* Unable to take oral medication reliably or have a malabsorption syndrome (i.e., 3 or more loose stools/day for at least 4 weeks associated with an unintentional weight loss of = or > 10 percent of body weight).
* History of sensitivity to the study medications.

Concurrent Medication:

Excluded:

* Maintenance therapy for opportunistic infections with macrolides or sulfonamides, immunomodulators, rifampin, amphotericin, dapsone, ganciclovir, antifolates, probenecid, benzodiazepines, nephrotoxins, and experimental cytotoxic chemotherapy.
* Medications such as aspirin, benzodiazepines, cimetidine, indomethacin, morphine, and sulfonamides should be avoided.

Concurrent Treatment:

Excluded:

* Lymphocyte replacement.

Patients with the following are excluded:

* Any medical or social condition that, in the opinion of the investigator, would adversely affect either participation or compliance in the study.
* Diagnosis of AIDS and febrile and have evidence of another serious opportunistic infection or central nervous system impairment.

Prior Medication:

Excluded:

* Maintenance therapy for opportunistic infections with macrolides or sulfonamides, immunomodulators, rifampin, amphotericin, dapsone, ganciclovir, antifolates, probenecid, benzodiazepines, nephrotoxins, and experimental cytotoxic chemotherapy within past 14 days.

Prior Treatment:

Excluded:

* Lymphocyte replacement within past 14 days.

Patients have the following symptoms and conditions:

* Laboratory evidence of HIV infection.
* Serological evidence of exposure to Toxoplasma gondii, but no clinical evidence of active toxoplasmic infection.
* Able to understand and sign a written informed consent.
* Either homosexual male or intravenous drug user.

Required:

* Stable prescribed dose of zidovudine (AZT) of at least 500 mg/day for 4 weeks.

Intravenous drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Study Completion 1995-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B Luft, Study Chair
Locations (2):
- United States (2):
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina

REFERENCES:
- [Background] Jacobson JM, Davidian M, Rainey PM, Hafner R, Raasch RH, Luft BJ. Pyrimethamine pharmacokinetics in human immunodeficiency virus-positive patients seropositive for Toxoplasma gondii. Antimicrob Agents Chemother. 1996 Jun;40(6):1360-5. doi: 10.1128/AAC.40.6.1360. PMID 8726001